CLINICAL TRIAL: NCT00169702
Title: The Effect of a Weight Management Program to Prevent Weight Gain and Metabolic Abnormalities During Treatment With the Atypical Neuroleptic Olanzapine: A Randomised Study
Brief Title: The Effect of a Weight Management Program During Treatment With Olanzapine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Eli Lilly and Company (Industry); Else Kröner-Fresenius-Centre for Nutritional Medicine (Unknown); Technical University of Munich (Other)
Responsible Party: Cordes, Joachim, Heinrich-Heine University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F1D-SB-018
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2007-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, weight management programme
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Other): standard information
  Interventions: Behavioral: weight management program
- Intervention (Active Comparator): weight management program, 12 sessions, 2 weekly, psychoeducational program, interactive topics like healthy food, diet behavior, physical activity, stress reduction.
  Interventions: Behavioral: weight management program

INTERVENTIONS:
Behavioral: weight management program — 12 sessions, psychoeducation
Behavioral: weight management program — 2 weekly, 12 sessions, psychoeducational weight management
  Arms: Standard

SUMMARY:
The study is a prospective, randomized, open-label study.

DETAILED DESCRIPTION:
The principal objective of this trial is to investigate the effect of a comprehensive behavioural treatment program on weight gain in schizophrenic patients under olanzapine treatment, and on subjective well-being.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for schizophrenia
* Ages between 18 and 65
* Informed consent
* Weight gain of at least 1.5 kg in the first 4 weeks
* A sufficient understanding to participate adequately in the weight management program
* Patients must agree to cooperate with all tests and examinations required by the protocol.
* Each patient must understand the nature of the study and must sign an informed consent document.

Exclusion Criteria:

* Serious, unstable somatic illnesses
* Illnesses associated with weight gain including renal and endocrine diseases
* Weight change greater than 3 kg in the preceding three months
* Weight gain less than 1.5 kg in the first 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-06; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
difference in mean weight gain | November 2007

SECONDARY OUTCOMES:
changes in waist circumference, blood pressure, blood lipids, fasting glucose | November 2007

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Cordes, MD, Principal Investigator — Department of Psychiatry and Psychotherapy at the Heinrich-Heine-University Düsseldorf, Rhineland State Clinics Düsseldorf, Bergische Landstrasse 2, 40629 Düsseldorf, Germany; Ansgar Klimke, Prof, Study Director — Department of Psychiatry, Offenbach; Hans Hauner, Prof, Study Director — Technical University of Munic
Locations (1):
- Heinrich-Heine-University, Rhineland State Clinics Düsseldorf, Düsseldorf, Rhineland State, Germany

REFERENCES:
- [Background] Hauner H, Rohrig K, Hebebrand J, Skurk T. No evidence for a direct effect of clozapine on fat-cell formation and production of leptin and other fat-cell-derived factors. Mol Psychiatry. 2003 Mar;8(3):258-9. doi: 10.1038/sj.mp.4001246. No abstract available. PMID 12660797